CLINICAL TRIAL: NCT03752970
Title: Mechanism of Action and Clinical Effect of BI 655130 in Patients With Fistulizing Crohn's Disease
Brief Title: A Study Testing How BI 655130 Works in Patients With Fistulizing Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1368-0008; 2017-003090-34 (EudraCT Number)
Record Dates: First submitted 2018-11-22; First posted 2018-11-26 (Actual); Results first posted 2024-02-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — spesolimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Screening Cohort (No Intervention): Patients enrolled in the Screening Cohort did not receive study treatment. This was a feasibility phase for fistula preparation and seton placement to determine the tissue samples that were suitable for analysis of the primary endpoint in the Study Cohort.
- Study Cohort - Placebo (Placebo Comparator): Patients with perianal fistulising Crohn's disease received Placebo intravenously every 4 weeks (week 0, 4, 8). At week 12 achievement of combined perianal fistula remission was determined, patients without combined perianal fistula remission were switched to spesolimab and were treated with spesolimab 1200 milligram intravenously every 4 weeks (week 12, 16 and 20). Patients with combined perianal fistula remission remained on Placebo and were treated with placebo intravenously every 4 weeks (week 12, 16 and 20).
  Interventions: Drug: Spesolimab; Drug: Placebo
- Study Cohort - Spesolimab (Experimental): Patients with perianal fistulising Crohn's disease received Spesolimab 1200 milligram intravenously every 4 weeks (week 0, 4, 8, 12, 16 and 20). At week 12 Placebo patients without combined perianal fistula remission were switched to spesolimab and were treated with spesolimab 1200 milligram intravenously every 4 weeks (week 12, 16 and 20).
  Interventions: Drug: Spesolimab

INTERVENTIONS:
Drug: Spesolimab — Spesolimab 1200 milligram intravenously every 4 weeks (week 0, 4, 8, 12, 16 and 20). At week 12 Placebo patients without combined perianal fistula remission were switched to spesolimab and were treated with spesolimab 1200 milligram intravenously every 4 weeks (week 12, 16 and 20).
  Arms: Study Cohort - Placebo; Study Cohort - Spesolimab
Drug: Placebo — Placebo intravenously every 4 weeks (week 0, 4, 8). At week 12 achievement of combined perianal fistula remission was determined, patients without combined perianal fistula remission were switched to spesolimab and were treated with spesolimab 1200 milligram intravenously every 4 weeks (week 12, 16 and 20). Patients with combined perianal fistula remission remained on Placebo and were treated with placebo intravenously every 4 weeks (week 12, 16 and 20).
  Arms: Study Cohort - Placebo

SUMMARY:
This is a study in adults with Crohn's Disease who also have fistulas near the anus. The study has 2 parts. The first part is to find out more about what causes the fistulas. In this part of the study, tissue samples are taken from patients. The second part of the study tests whether a medicine called spesolimab (BI 655130) helps patients with Crohn's Disease.

Participants get study medication for 24 weeks. The participants are put into 2 groups. It is decided by chance who gets into which group. One group gets an intravenous drip that contains spesolimab every 4 weeks. The other group gets a placebo drip every 4 weeks. The placebo drip looks like the spesolimab drip, but contains no medicine.

The doctors regularly examine fistulas of the participants. The results of the fistula examinations are compared between the groups. The doctors also check the general health of the patients.

ELIGIBILITY:
Inclusion criteria

* 18-75 years at date of signing informed consent
* Male or female patients. Women of childbearing potential (WOCBP)1 must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. Restrictions regarding women of childbearing potential. Restrictions regarding contraception for female patients are not applicable for Screening Cohort
* Diagnosis of clinical Crohn´s Disease ≥ 3 months prior to screening by clinical and endoscopic evidence and corroborated by a histopathology report
* Has ≥ 1 perianal active* fistula(s) with clinical indication for seton drainage (≥ 4 weeks duration before enrolment, as a complication of CD) **

  * Criteria for Active Fistula: As per clinical evaluation: Presence of spontaneous drainage or drainage after gentle finger compression at the external openings & as confirmed by radiological (MRI) exploration

  ** Patients who are screened with a seton drainage in place are eligible provided the drainage has not been in place for > 3 months and the patient meets the rest of the eligibility criteria
* Absent, mild or moderate clinical activity with CDAI < 250. CDAI is not applicable for Screening Cohort
* Demonstrated in the past inadequate fistula response or loss of response or have had unacceptable side effects with approved doses of at least one of the following compounds: immunosuppressive agents (e.g. thiopurines, methotrexate), TNFɑ antagonists (e.g. infliximab, adalimumab, certolizumab pegol; or respective biosimilars), vedolizumab, ustekinumab, azathioprine and / or antibiotics
* Patients with family history of colorectal cancer or personal history of increased colorectal cancer risk must have had a negative ileocolorectal cancer screening within <1 year prior to screening per local guidance
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
* Further inclusion criteria apply

Gastrointestinal Exclusion Criteria (Study cohort only)

* Complications of Crohn's Disease such as symptomatic strictures, functional stenosis distal from fistula(s), short gut syndrome, or any other manifestation that might require surgery, could preclude the use of the PDAI and CDAI to assess response to therapy, or would possibly confound the evaluation of benefit from treatment with BI 655130
* Rectovaginal fistulas
* Anticipated to require surgical intervention for CD including any fistula surgical procedures (except seton drainage)
* Has an abscess that the investigator feels requires drainage beyond fistula drainage with a seton (based on either clinical assessment or MRI)
* Any kind of bowel resection or diversion within 6 months or any other intraabdominal surgery within 3 months prior to screening.
* Ileostomy, colostomy or known fixed symptomatic stenosis of the intestine at screening
* Positive stool examinations for C. difficile or other intestinal pathogens < 30 days prior to screening

  -- Evidence of colonic mucosal dysplasia or colonic adenomas, unless properly removed (properly according to the investigator's assessment)
* Faecal Microbiota transplant (FMT) within 6 months prior to randomization
* Treatment with:

  * any non-biologic medication (incl. cyclosporine, JAK inhibitors such as tofacitinib, tacrolimus, sirolimus, mycophenolate mofetile, S1P modulators, SMAD7 antisense inhibitors such as mongersen), other than those allowed per chapter 4.2.1 within 30 days prior to randomisation unless these patients show an undetectable plasma concentration
  * any biologic treatment approved for CD other than anti-TNFα inhibitors within 8 weeks prior to randomization unless these patients show an undetectable plasma concentration
  * any investigational or non-approved biologic for CD (including but not limited to IL-23 inhibitors) within 12 weeks prior to randomisation or etrolizumab within 8 weeks prior to randomization unless these patients show an undetectable plasma concentration
  * rectal 5-ASA, rectal Tacrolimus, parenteral or rectal corticosteroids (incl. budesonide) within 2 weeks prior to randomisation
  * any antibiotics within 1 week prior to randomisation
  * any prior autologous or allogeneic, haematopoietic (HSC) or mesenchymal stem cell (MSC) therapy
  * any prior exposure to BI 655130
  * any chronic use of NSAID within 2 weeks prior to randomisation (occasional use of NSAIDs and acetaminophen for headache, arthritis, myalgias, menstrual cramps, etc., and daily use of baby or low dose (81-162.5mg) aspirin for cardiovascular prophylaxis are permitted)
  * any life-attenuated vaccines within 6 weeks prior to randomization

Infectious Disease Exclusion Criteria (Study cohort only)

* Increased risk of infectious complications (e.g. due to past organ or stem cell transplantation)
* Live or attenuated vaccination within 6 weeks prior to randomization
* Patients with a positive QuantiFERON TB test during screening are excluded, unless:

  * Patient had previous diagnosis of active or latent TB and has completed appropriate treatment per local practice/guidelines within the last 3 years and at least 6 months before first administration of trial medication under this protocol (patients may be re-screened once to meet this criterion)
  * Patients with suspected false positive or indeterminate QuantiFERON TB result may be re-tested once
  * If Quantiferon not available or providing indeterminate results after repeat testing : A tuberculin skin test reaction ≥10mm (≥5mm if receiving ≥15mg/d prednisone or its equivalent)
* Relevant chronic or acute infections including active tuberculosis, human immunodeficiency virus (HIV) infection or viral hepatitis. A patient can be re-screened if the patient was treated and is cured from the acute infection.

General Exclusion Criteria (Study cohort only)

* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ carcinoma of uterine cervix.
* Major surgery (major according to the investigator's assessment) performed within 12 weeks prior to randomization or planned during study conduct, e.g. hip replacement.
* Pathological safety lab parameters: haemoglobin < 8 g/dL, total white blood count (WBC) < 3000 cells/μl, neutrophils < 1000 cells/μl, thrombocytes < 100.000/μl, creatinine ≥ 2 mg/dL, total bilirubin > 2 x ULN with ratio of direct/indirect >1 (patients with Gilbert's syndrome are not excluded), Alkaline Phosphatase >3 x ULN.
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Previous enrolment in this trial (exception: patients of screening cohort may be enrolled in study cohort)
* Currently enrolled in another investigational device or drug trial
* Women who are pregnant, nursing, or who plan to become pregnant in the trial
* Evidence of a current or previous disease, medical condition (including chronic alcohol or drug abuse) other than Crohn´s disease, surgical procedure, medical examination finding (including vital signs and electrocardiogram (ECG)), or laboratory value at the screening visit outside the reference range that in the opinion of the investigator is clinically significant and would make the study participant unreliable to adhere to the protocol or to complete the trial, compromise the safety of the patient, or compromise the quality of the data
* History of allergy/hypersensitivity to the systemically administered trial medication agent or its excipients or to contrast media

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-07-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- AKH - Medical University of Vienna, Vienna, Austria
- Belgium (2):
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Herlev and Gentofte Hospital, Herlev, Denmark
- Germany (2):
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Ulm, Ulm
- Semmelweis University, Budapest, Hungary
- Amsterdam UMC, Locatie AMC, Amsterdam, Netherlands
- Inje University Haeundae Paik Hospital, Busan, South Korea
- Hospital Universitari de Girona Doctor Josep Trueta, Girona, Spain

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Lebwohl MG, Thoma C, Haeufel T. Spesolimab use in generalised pustular psoriasis flares - Authors' reply. Lancet. 2024 Aug 31;404(10455):847-848. doi: 10.1016/S0140-6736(24)01557-5. No abstract available. PMID 39216969
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was divided into a Screening Cohort and a Study Cohort:
  Screening Cohort did not receive study treatment.
  Study Cohort was a randomised, double-blind, placebo-controlled, Phase IIa design, and was conducted in 2 periods each of 12 weeks' duration. Patients who completed Week 24 of Period 2 and had clinical benefit were offered continued treatment in an open label, long-term extension study. Patients who did not continue into the extension study were followed up at Week 36.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Screening Cohort
Arm/Group | Screening Cohort | Study Cohort - Placebo | Study Cohort - Spesolimab
Started | 6 | 0 | 0
Completed | 6 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Study Cohort Period 1 (Week 1 - <week12)
Arm/Group | Screening Cohort | Study Cohort - Placebo | Study Cohort - Spesolimab
Started (Subjects in the screening and study cohorts are mutually exclusive.) | 0 | 10 | 11
Completed | 0 | 9 | 9
Not Completed | 0 | 1 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Study Cohort Week 12 Assignment
Arm/Group | Screening Cohort | Study Cohort - Placebo | Study Cohort - Spesolimab
Started | 0 | 9 | 9
Switching Patients (Patients switching to Spesolimab) | 0 | 4 (Patients switching to Spesolimab in period 2) | 0
Completed | 0 | 5 (Patients staying on Placebo in period 2) | 9
Not Completed | 0 | 4 | 0
Not completed — Switched to Spesolimab in period 2 | 0 | 4 | 0
Period: Study Cohort - Period 2 (>=Week 12 - 24)
Arm/Group | Screening Cohort | Study Cohort - Placebo | Study Cohort - Spesolimab
Started | 0 | 5 | 13 (Combination of period 1 Spesolimab patients and period 1 Placebo subjects who switched to Spesolimab in period 2.)
Completed | 0 | 5 | 12
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects who entered the Screening Cohort or the Study Cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Screening Cohort | Study Cohort - Placebo | Study Cohort - Spesolimab | Total
Number analyzed (Participants) | 6 | 10 | 11 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (10.8) | 34.0 (8.3) | 39.2 (10.8) | 38.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 9
  Male | 2 | 7 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 10 | 11 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 6 | 8 | 10 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Total Number of Deregulated Genes at Week 4
Description: The total number of deregulated genes based on biopsies from the inner fistula orifice at Week 4 comparing changes in gene expression from baseline between the two treatment groups. For each gene, a repeated measures linear regression model was utilized with treatment (BI 655130 or Placebo), visit (baseline, week 4), treatment by visit interaction as fixed effect and patient as a blocking factor.
  Changes will be quantified by log2 fold changes (FC) and associated False Discovery Rate (FDR) adjusted p-values.
  Genes will be considered deregulated if they fulfil the following criteria:
  * FDR adjusted p-value ≤ 0.05
  * |fold change| ≥ 1.5 (|log2 fold change| ≥ 0.58)
Time Frame: Biopsies taken at screening (Week -3) and at week 4 of treatment.
Population: RNA Sequencing Set: All patients who were randomised and treated with any amount of study drug and who provide a valid baseline and at least one valid post-baseline observation for at least one gene expression variable of biopsy. Data analysed with original results (OR) approach, implying the presentation of data exactly as observed.
Measure: Number; unit: Deregulated genes
Arm/Group | Study Cohort - Placebo | Study Cohort - Spesolimab
Number analyzed (Participants) | 9 | 7
Deregulated genes | 0 | 0

2. Secondary Outcome: Number of Patients With Perianal Fistula Response at Week 12
Description: Number of patients with perianal fistula response at Week 12 defined as closure of at least 50% of external openings, no drainage/discharge despite gentle finger compression of fistulas that were draining at baseline and without new emerging fistulas.
  The no response imputation (NRI) approach is applied: missing visits where imputed whereby all subsequent visits after a patient took rescue medication for the disease under study or died due to any cause were considered to be missing.
Time Frame: At baseline (day 1) and week 12 (day 85) of treatment.
Population: Includes all patients of the Study Cohort who provided a baseline value and at least one post-baseline value for at least one secondary endpoint or further efficacy endpoint. Following the intent-to-treat principle, patients will be analysed according to the treatment they were assigned to at randomisation.
Measure: Number; unit: Participants
Arm/Group | Study Cohort - Placebo | Study Cohort - Spesolimab
Number analyzed (Participants) | 10 | 11
Participants | 7 | 1
Statistical Analysis 1: Comparison: Study Cohort - Placebo vs Study Cohort - Spesolimab; Test type: Other; Risk Difference (RD) = -0.609, 95% CI 2-sided [-0.880 to -0.186]

3. Secondary Outcome: Number of Patients With Perianal Fistula Remission at Week 12
Description: Proportion of patients with perianal fistula remission at Week 12 defined as closure of all external openings, no drainage/discharge despite gentle finger compression of fistulas that were draining at baseline and without new emerging fistulas.
  The no response imputation (NRI) approach is applied: missing visits where imputed whereby all subsequent visits after a patient took rescue medication for the disease under study or died due to any cause were considered to be missing.
Time Frame: At baseline (day 1) and week 12 (day 85) of treatment.
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Study Cohort - Placebo | Study Cohort - Spesolimab
Number analyzed (Participants) | 10 | 11
Participants | 6 | 1
Statistical Analysis 1: Comparison: Study Cohort - Placebo vs Study Cohort - Spesolimab; Test type: Other; Risk Difference (RD) = -0.509, 95% CI 2-sided [-0.816 to -0.087]

4. Secondary Outcome: Number of Patients With Combined Perianal Fistula Remission at Week 12
Description: Number of patients with combined perianal fistula remission at Week 12 defined as closure of all external openings, no drainage/discharge despite gentle finger compression of fistulas that were draining at baseline and without new emerging fistulas, AND absence collections of >2 centimeter, confirmed by magnetic resonance imaging (MRI) in at least 2 of 3 dimensions - blinded and centrally read.
  The no response imputation (NRI) approach is applied: missing visits where imputed whereby all subsequent visits after a patient took rescue medication for the disease under study or died due to any cause were considered to be missing.
Time Frame: At baseline (day 1) and week 12 (day 85) of treatment.
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Study Cohort - Placebo | Study Cohort - Spesolimab
Number analyzed (Participants) | 10 | 11
Participants | 6 | 1
Statistical Analysis 1: Comparison: Study Cohort - Placebo vs Study Cohort - Spesolimab; Test type: Other; Risk Difference (RD) = -0.509, 95% CI 2-sided [-0.816 to -0.087]

ADVERSE EVENTS:
Time Frame: Screening cohort: up to 56 days. Period 1: From start of treatment (Placebo or Spesolimab) in period 1 till start of treatment (Placebo or Spesolimab) in period 2, up to 84 days. Period 2: From start of treatment (Placebo or Spesolimab) in period 2 till end of last infusion (Placebo or Spesolimab) in period 2 + residual effect period of 112 days, up to 182 days.
Description: Screening cohort: all patients of the Screening Cohort who entered the trial.
  Study cohort: all patients who were randomised and treated with any amount of study drug.
Groups:
- Study Cohort Period 1: Placebo: Patients with perianal fistulising Crohn's disease received Placebo intravenously every 4 weeks (week 0, 4, 8). The arm only considers adverse events reported in period 1.
- Study Cohort Period 1: Spesolimab: Patients with perianal fistulising Crohn's disease received Spesolimab 1200 milligram intravenously every 4 weeks (week 0, 4, 8). The arm only considers adverse events reported in period 1.
- Study Cohort Period 2: Placebo - Placebo: Patients with perianal fistulising Crohn's disease received Placebo intravenously every 4 weeks (week 0, 4, 8, 12, 16 and 20). The arm only considers adverse events reported in period 2.
- Study Cohort Period 2: Placebo - Spesolimab: Patients with perianal fistulising Crohn's disease received Placebo intravenously every 4 weeks (week 0, 4, 8). At week 12 achievement of combined perianal fistula remission was determined, patients without combined perianal fistula remission were switched to spesolimab and were treated with spesolimab 1200 milligram intravenously every 4 weeks (week 12, 16 and 20). The arm only considers adverse events reported in period 2.
- Study Cohort Period 2: Spesolimab - Spesolimab: Patients with perianal fistulising Crohn's disease received Spesolimab 1200 milligram intravenously every 4 weeks (week 0, 4, 8, 12, 16 and 20). The arm only considers adverse events reported in period 2.
Arm/Group | Screening Cohort | Study Cohort Period 1: Placebo | Study Cohort Period 1: Spesolimab | Study Cohort Period 2: Placebo - Placebo | Study Cohort Period 2: Placebo - Spesolimab | Study Cohort Period 2: Spesolimab - Spesolimab
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/10 | 0/11 | 0/5 | 0/4 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/10 | 1/11 | 1/5 | 0/4 | 0/9
Other Adverse Events (participants affected / at risk) | 1/6 | 9/10 | 6/11 | 3/5 | 4/4 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Screening Cohort (N=6) | Study Cohort Period 1: Placebo (N=10) | Study Cohort Period 1: Spesolimab (N=11) | Study Cohort Period 2: Placebo - Placebo (N=5) | Study Cohort Period 2: Placebo - Spesolimab (N=4) | Study Cohort Period 2: Spesolimab - Spesolimab (N=9)
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Screening Cohort (N=6) | Study Cohort Period 1: Placebo (N=10) | Study Cohort Period 1: Spesolimab (N=11) | Study Cohort Period 2: Placebo - Placebo (N=5) | Study Cohort Period 2: Placebo - Spesolimab (N=4) | Study Cohort Period 2: Spesolimab - Spesolimab (N=9)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Enanthema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Asymptomatic COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Latent tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 3 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
For the primary endpoint, due to the limited number of evaluable samples from the curettage at baseline and at Week 4, curettage biopsies were not included in the gene expression analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT03752970/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT03752970/SAP_001.pdf